CLINICAL TRIAL: NCT02139176
Title: Assessing Strategies for Increasing Male Involvement in Malawi's Antenatal Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-3707
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2016-09

CONDITIONS: HIV
Keywords: couple HIV testing and counseling; disclosure; discordant; HIV; Malawi
MeSH Terms: interventions — Contact Tracing; Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient referral (Active Comparator): Women are given an invitation to give to a male partner inviting them to come to the clinic for important pregnancy information
  Interventions: Behavioral: patient referral
- contract referral (Experimental): Same as control. However, if the male partner does not present, a community worker will trace the partner in the community.
  Interventions: Behavioral: contract referral; Behavioral: patient referral

INTERVENTIONS:
Behavioral: contract referral — A female partner signs a contract saying it is permissible for a community worker to trace a male sex partner in the community.
  Other Names: partner notification; contract partner notification; invitation plus tracing
  Arms: contract referral
Behavioral: patient referral — A patient agrees to recruit their partner using the invitation.
  Other Names: passive referral; patient notification; invitation only

SUMMARY:
In sub-Saharan Africa, engaging men in HIV prevention, care, and treatment has proven challenging. Along all steps of the HIV care-seeking cascade, men exhibit worse care-seeking behaviors than women. They are less likely to be tested for HIV, initiate combination antiretroviral therapy (cART), and be retained in cART care. Additionally, men rarely engage in the care of their female sex partners, even though couple care-seeking is associated with marked improvements in condom use within HIV-discordant couples. Option B+, Malawi's program for providing immediate, lifelong combination antiretroviral therapy (cART) to all HIV-infected pregnant women at the time of diagnosis, is an important entry-point for involving male partners in care.

This is a pilot randomized controlled trial (N=200 women) comparing two strategies of male partner involvement within the Option B+ program. In both arms (patient referral and contract referral) women will be encouraged to invite their male partners to accompany them to the clinic for couple HIV counseling and testing. In the contract referral arm, if the couple does not present within one week, the male partner will receive a home visit encouraging them to present to the clinic. We will compare the two arms for 1) uptake of couple HIV counseling and testing (cHCT), 2) uptake of cART for women, and 3) linkage to care for HIV-infected men. Results are expected to inform a larger trial and ultimately improve care-seeking in Malawi's HIV program.

Objective 1: Determine acceptability of male partner recruitment for cHTC within an Option B+ context. We will assess acceptability of eligible females to participate in this pilot RCT and reasons for non-participation.

Objective 2: Assess whether study arm (patient referral versus contract referral) is associated with cHTC uptake. We will conduct a pilot randomized controlled trial (RCT) of male partner recruitment. This study will contain two arms: patient referral and contract referral for uptake of cHTC (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or 16-17 years old and married

  * Pregnant
  * Received a positive HIV-test within the last day
  * Will be in Lilongwe for the next month
  * Able and willing to give locator information for >1 male partner in the Bwaila District Hospital catchment area (either a mobile number, a physical address, or both)

Exclusion Criteria:

* Enrolled/enrolling in the PROMISE study
* Initially Presenting with a male sex partner

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nora E Rosenberg, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Mina Hosseinipour, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bwaila District Hospital Antenatal Unit, Lilongwe, Central District, Malawi

REFERENCES:
- [Derived] Rosenberg NE, Mtande TK, Saidi F, Stanley C, Jere E, Paile L, Kumwenda K, Mofolo I, Ng'ambi W, Miller WC, Hoffman I, Hosseinipour M. Recruiting male partners for couple HIV testing and counselling in Malawi's option B+ programme: an unblinded randomised controlled trial. Lancet HIV. 2015 Nov;2(11):e483-91. doi: 10.1016/S2352-3018(15)00182-4. Epub 2015 Oct 22. PMID 26520928

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Referral | Contract Referral
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: HIV-infected women eligible for Option B+
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Referral | Contract Referral | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (0.49) | 26.6 (0.50) | 26.6 (0.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Who Came With Their Partners and Received Couple Counseling and Testing
Description: Based on whether the female partner brings her male partner to the antenatal clinic for couple HIV counseling and testing (as recorded on study case report forms) as the primary measure of uptake. We will compare time to couple HIV counseling and testing between groups using the Kaplan Meier method and a log rank test.
Time Frame: three months
Measure: Number; unit: Female participants receiving CHTC
Arm/Group | Patient Referral | Contract Referral
Number analyzed (Participants) | 100 | 100
Female participants receiving CHTC | 52 | 70

2. Secondary Outcome: Female First Option B+ Follow-up Visit
Description: It will be assessed whether the female participants return for their first Option B+ visit (using the clinic's routine Option B+ records). The number retained will be compared.
Time Frame: three months
Measure: Number; unit: participants
Arm/Group | Patient Referral | Contract Referral
Number analyzed (Participants) | 100 | 100
participants | 83 | 91

3. Secondary Outcome: Male Linkage to Care
Description: It will be assessed whether newly diagnosed HIV-infected male partners are linked to care within one month of learning their HIV positive result with their partner. This will be assessed from abstraction of routine clinic records at Martin Preuss Center.
Time Frame: one month from male presentation to the clinic
Population: These are only the HIV-infected men who participated in the study who were HIV-infected and not already engaged in care. That is why it is only a subset of the larger population.
Measure: Number; unit: partners linked to care
Arm/Group | Patient Referral | Contract Referral
Number analyzed (Participants) | 26 | 33
partners linked to care | 5 | 15

ADVERSE EVENTS:
Arm/Group | Patient Referral | Contract Referral
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 3/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Referral (N=100) | Contract Referral (N=100)
social disruptions reported by women (Social circumstances) | 0 (0) | 3 (3) — * Two couples separated and the woman reported this * One female participant felt blamed for bringing HIV into the relationship and she reported this * One male participant was upset when he misunderstood which partner he was being called about.
social disruption reported by men (Social circumstances) | 0 (0) | 1 (1) — Men who reported disruptions related to tracing or study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No